CLINICAL TRIAL: NCT01466582
Title: Comorbidity and Aging With HIV, the agehIV Cohort Study
Brief Title: Comorbidity and Aging With HIV
Acronym: agehIV
Status: Active, not recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Public Health Service of Amsterdam (Other Government)
Responsible Party: Principal Investigator, Prof. dr. Peter Reiss, Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL30802.018.09
Record Dates: First submitted 2011-10-31; First posted 2011-11-08 (Estimated); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: HIV-1-infection; Comorbidity; Ageing
Keywords: HIV-1-infection; comorbidity; ageing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum (EDTA/heparin/citrate), PBMCs, urine, stool (for future microbiome studies)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-negative controls: A group of HIV-negative controls, aged 45 years and above, that is recruited at the STD-clinic of the Public Health Service Amsterdam or at the existing Amsterdam Cohort Studies.
- HIV-positive patients: A group of HIV-1-infected patients, aged 45 years and above, that is recruited at the HIV outpatient clinic of the Academic Medical Center.

SUMMARY:
In this prospective cohort study the investigators will assess the prevalence and incidence of a broad range of age-related co-morbidities and their (known) risk factor among HIV-patients and HIV-negative controls. HIV might cause premature onset or accelerated aging and could therefore result in an increase of age-related comorbidities when compared with controls.

DETAILED DESCRIPTION:
The standard use of combination antiretroviral therapy (cART) has resulted in major and sustained declines in HIV-associated morbidity and mortality. Nonetheless, the life expectancy of patients with HIV on cART still remains 10 or more years shorter than that of uninfected persons of the same age, especially in patients starting cART at the time infection is already advanced. A greater risk of a broad range of co-morbidities, experienced by as many as 60% of patients, even after adjustment for age, may contribute to this discrepancy. Several studies have demonstrated an increased incidence of heart disease, diabetes mellitus, kidney disease, liver disease, osteoporosis, malignancies (other than Kaposi's sarcoma and non-Hodgkin's lymphoma traditionally associated with HIV), cognitive disorders and possibly chronic obstructive pulmonary disease in HIV-infected individuals when compared to age matched HIV-uninfected controls. Of note, the incidence of each of the mentioned co-morbidities is also higher after adjustment for age and other traditional risk factors. Most studies were conducted in the United States where prevalence of and risk factors for the various co-morbidities may be different than in Europe, in particular the Netherlands.

HIV-related factors and adverse effects of cART each may independently contribute to the observed increased risk of several of the earlier mentioned co-morbidities. Interestingly, HIV-infected men in the absence of cART have increased frailty (a clinical syndrome associated with aging that identifies a subset of older adults at high risk of mortality and other adverse outcomes) when compared to uninfected men of similar age. Middle aged HIV-infected men despite cART use also show reduction in exercise capacity, functional performance, physical activity, and grip strength.

The multidisciplinary expertise regarding co-morbidities which is present within the AMC in close collaboration with the existing data collection structures of the HIV Monitoring Foundation (HMF) and the Cluster of Infectious Diseases of the Public Health Service Amsterdam (PHSA), offers a unique opportunity to systematically identify the burden of co-morbidity, their (known) risk factors and their effect on quality of life among HIV-infected individuals and in a comparable group of uninfected individuals.

As of August 2020, the study was amended to include a substudy, the main aim of which is to determine and compare the rate of SARS-CoV-2 infection, the extent of the SARS-CoV-2-specific adaptive immune response, and the incidence and severity of COVID-19 disease between PWH and HIV-negative cohort participants who remain in active follow-up.

Furthermore, if disease prevalence is sufficiently high, another aim will be to determine and compare risk factors for the development of severe COVID-19 between PWH and HIV-negative controls. Furthermore, an attempt will be made to compare the impact of nationally imposed social distancing measures on substance use, medication adherence, sexual behavior, quality of life and depressive symptoms in study participants.

Specific aims

1. To assess the SARS-CoV-2 infection rate in HIV-positive and -negative participants over 24 months by combined testing for in vivo SARS-CoV-2 specific antibodies, and in vitro SARS-CoV-2 specific memory B-cell and T-cell responses.
2. To assess the course over time of SARS-CoV-2 specific antibody levels, the quantity of SARS-CoV-2-specific memory B-cell, as well as CD4 and CD8 T-cell responses, and the functionality of the overall T cell response in vitro in HIV-positive and -negative participants with demonstrated SARS-CoV-2 infection, as well as the presence of SARS-CoV-2 cross-reactive common cold coronavirus (HKU1, OC43, NL63 and 229E) specific CD4 and CD8 T-cell responses in selected participants.
3. To assess the proportion of HIV-positive and -negative participants who carried broadly recognizing coronavirus (HKU1, OC43, NL63 and 229E) antibodies, prior to demonstrated SARS-CoV-2 infection.
4. To assess the rate and severity of COVID-19 disease in HIV-positive and -negative participants.
5. To assess factors associated with SARS-CoV-2 infection, development of COVID-19 and severe disease (i.e. requiring hospitalization and/or ICU-admission) in HIV-positive and HIV-negative participants.
6. To assess associations between nationally imposed social distancing measures and substance use, medication adherence, social behavior, quality of life and depression in study participants.

ELIGIBILITY:
Inclusion Criteria:

* For the HIV-positive patients: HIV-1 infection and aged 45 years and above
* For the HIV-negative controls: HIV-uninfected and aged 45 years and above

Exclusion Criteria:

* None

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The HIV-positive patients are recruited at the HIV outpatient clinic of the Academic Medical Center The HIV-negative controls are recruited at the STD-clinic of the Public Health Service Amsterdam and at the existing Amsterdam Cohort Studies.
Sampling Method: Non-Probability Sample
Enrollment: 1148 (Actual)
Dates: Start 2010-10; Primary Completion 2040-10 (Estimated); Study Completion 2040-10 (Estimated)

PRIMARY OUTCOMES:
The prevalence of comorbidities, organ system dysfunction and their risk factors at time of enrolment | at enrolment and after every 2 years follow up. The Ethics Committee has approved for the study to continue without a set end-date, depending on continued funding.
  To assess the prevalence and incidence of comorbidities, organ system dysfunction and their risk factors over two years of follow-up in a cohort of HIV-infected individuals (mostly on antiretroviral therapy) and in a cohort of comparable but uninfected controls
The incidence of comorbidities, organ system dysfunction and their risk factors after two years of follow up | After every 2 years of follow up.The Ethics Committee has approved for the study to continue without a set end-date, depending on continued funding.
  To assess the incidence of comorbidities, organ system dysfunction and their risk factors after tow years of follow up in a cohort of HIV-infected individuals (mostly on antiretroviral therapy) in comparison to that of a cohort of comparable but uninfected controls

SECONDARY OUTCOMES:
Quality of life measured using the Medical Outcomes Study Short Form 36-item health survey (SF-36) | At baseline and after 2 years
  To compare quality of life both at baseline and over time, between patients who are HIV-infected or HIV-uninfected, and with and without co-morbidity.
Management strategies | After 4 years
  To suggest appropriate management strategies for identified co-morbidities in the HIV-infected cohort and their risk factors, if advice is requested by the patient's HIV physician. To assess over time if the prevalence and incidence of co-morbidity burden have changed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Reiss, MD, PhD, Principal Investigator — Amsterdam University Medical Centers, University of Amsterdam, Amsterdam; Amsterdam Institute for Global Health and Development, Amsterdam; Maria Prins, PhD, Principal Investigator — Public Health Service Amsterdam, Amsterdam; Academic Medical Center, Amsterdam
Locations (2):
- Netherlands (2):
  - Public Health Service Amsterdam, Amsterdam
  - Academic Medical Center, Amsterdam

REFERENCES:
- [Background] Kooij KW, Vogt L, Wit FWNM, van der Valk M, van Zoest RA, Goorhuis A, Prins M, Post FA, Reiss P; AGEhIV Cohort Study. Higher Prevalence and Faster Progression of Chronic Kidney Disease in Human Immunodeficiency Virus-Infected Middle-Aged Individuals Compared With Human Immunodeficiency Virus-Uninfected Controls. J Infect Dis. 2017 Sep 15;216(6):622-631. doi: 10.1093/infdis/jix202. PMID 28934420
- [Background] van Zoest RA, van der Valk M, Wit FW, Vaartjes I, Kooij KW, Hovius JW, Prins M, Reiss P; AGEhIV Cohort Study Group. Suboptimal primary and secondary cardiovascular disease prevention in HIV-positive individuals on antiretroviral therapy. Eur J Prev Cardiol. 2017 Aug;24(12):1297-1307. doi: 10.1177/2047487317714350. Epub 2017 Jun 5. PMID 28578613
- [Background] Langebeek N, Kooij KW, Wit FW, Stolte IG, Sprangers MAG, Reiss P, Nieuwkerk PT; AGEhIV Cohort Study Group. Impact of comorbidity and ageing on health-related quality of life in HIV-positive and HIV-negative individuals. AIDS. 2017 Jun 19;31(10):1471-1481. doi: 10.1097/QAD.0000000000001511. PMID 28574965
- [Background] Su T, Mutsaerts HJ, Caan MW, Wit FW, Schouten J, Geurtsen GJ, Sharp DJ, Prins M, Richard E, Portegies P, Reiss P, Majoie CB; AGEhIV Cohort Study. Cerebral blood flow and cognitive function in HIV-infected men with sustained suppressed viremia on combination antiretroviral therapy. AIDS. 2017 Mar 27;31(6):847-856. doi: 10.1097/QAD.0000000000001414. PMID 28121708
- [Background] Kooij KW, Wit FW, Booiman T, van der Valk M, Schim van der Loeff MF, Kootstra NA, Reiss P; AGEhIV Cohort Study Group. Cigarette Smoking and Inflammation, Monocyte Activation, and Coagulation in HIV-Infected Individuals Receiving Antiretroviral Therapy, Compared With Uninfected Individuals. J Infect Dis. 2016 Dec 15;214(12):1817-1821. doi: 10.1093/infdis/jiw459. Epub 2016 Sep 28. PMID 27683822
- [Background] Kooij KW, Schouten J, Wit FW, van der Valk M, Kootstra NA, Stolte IG, van der Meer JT, Prins M, Grobbee DE, van den Born BJ, Reiss P. Difference in Aortic Stiffness Between Treated Middle-Aged HIV Type 1-Infected and Uninfected Individuals Largely Explained by Traditional Cardiovascular Risk Factors, With an Additional Contribution of Prior Advanced Immunodeficiency. J Acquir Immune Defic Syndr. 2016 Sep 1;73(1):55-62. doi: 10.1097/QAI.0000000000001024. PMID 27513572
- [Background] Su T, Wit FW, Caan MW, Schouten J, Prins M, Geurtsen GJ, Cole JH, Sharp DJ, Richard E, Reneman L, Portegies P, Reiss P, Majoie CB; AGEhIV Cohort Study. White matter hyperintensities in relation to cognition in HIV-infected men with sustained suppressed viral load on combination antiretroviral therapy. AIDS. 2016 Sep 24;30(15):2329-39. doi: 10.1097/QAD.0000000000001133. PMID 27149087
- [Background] van Zoest RA, Wit FW, Kooij KW, van der Valk M, Schouten J, Kootstra NA, Wiersinga WJ, Prins M, van den Born BJ, Reiss P; AGEhIV Cohort Study Group. Higher Prevalence of Hypertension in HIV-1-Infected Patients on Combination Antiretroviral Therapy Is Associated With Changes in Body Composition and Prior Stavudine Exposure. Clin Infect Dis. 2016 Jul 15;63(2):205-13. doi: 10.1093/cid/ciw285. Epub 2016 May 3. PMID 27143668
- [Background] Kooij KW, Wit FW, van Zoest RA, Schouten J, Kootstra NA, van Vugt M, Prins M, Reiss P, van der Valk M; AGEhIV Cohort Study Group. Liver fibrosis in HIV-infected individuals on long-term antiretroviral therapy: associated with immune activation, immunodeficiency and prior use of didanosine. AIDS. 2016 Jul 17;30(11):1771-80. doi: 10.1097/QAD.0000000000001119. PMID 27088320
- [Background] Cobos Jimenez V, Wit FW, Joerink M, Maurer I, Harskamp AM, Schouten J, Prins M, van Leeuwen EM, Booiman T, Deeks SG, Reiss P, Kootstra NA; AGEhIV Study Group. T-Cell Activation Independently Associates With Immune Senescence in HIV-Infected Recipients of Long-term Antiretroviral Treatment. J Infect Dis. 2016 Jul 15;214(2):216-25. doi: 10.1093/infdis/jiw146. Epub 2016 Apr 12. PMID 27073222
- [Background] Demirkaya N, Wit FW, van Den Berg TJ, Kooij KW, Prins M, Schlingemann RO, Abramoff MD, Reiss P, Verbraak FD; AGEhIV Cohort Study Group. HIV-Associated Neuroretinal Disorder in Patients With Well-Suppressed HIV-Infection: A Comparative Cohort Study. Invest Ophthalmol Vis Sci. 2016 Mar;57(3):1388-97. doi: 10.1167/iovs.15-18537. PMID 27018841
- [Background] Schouten J, Su T, Wit FW, Kootstra NA, Caan MW, Geurtsen GJ, Schmand BA, Stolte IG, Prins M, Majoie CB, Portegies P, Reiss P; AGEhIV Study Group. Determinants of reduced cognitive performance in HIV-1-infected middle-aged men on combination antiretroviral therapy. AIDS. 2016 Apr 24;30(7):1027-38. doi: 10.1097/QAD.0000000000001017. PMID 26752277
- [Background] Moller LM, Brands R, Sluiter JK, Schouten J, Wit FW, Reiss P, Prins M, Stolte IG. Prevalence and determinants of insufficient work ability in older HIV-positive and HIV-negative workers. Int Arch Occup Environ Health. 2016 May;89(4):699-709. doi: 10.1007/s00420-015-1108-0. Epub 2016 Jan 8. PMID 26747456
- [Background] Su T, Caan MW, Wit FW, Schouten J, Geurtsen GJ, Cole JH, Sharp DJ, Vos FM, Prins M, Portegies P, Reiss P, Majoie CB; AGEhIV Cohort Study. White matter structure alterations in HIV-1-infected men with sustained suppression of viraemia on treatment. AIDS. 2016 Jan;30(2):311-22. doi: 10.1097/QAD.0000000000000945. PMID 26691551
- [Background] Kooij KW, Wit FW, Schouten J, van der Valk M, Godfried MH, Stolte IG, Prins M, Falutz J, Reiss P; AGEhIV Cohort Study Group. HIV infection is independently associated with frailty in middle-aged HIV type 1-infected individuals compared with similar but uninfected controls. AIDS. 2016 Jan;30(2):241-50. doi: 10.1097/QAD.0000000000000910. PMID 26684821
- [Result] Su T, Schouten J, Geurtsen GJ, Wit FW, Stolte IG, Prins M, Portegies P, Caan MW, Reiss P, Majoie CB, Schmand BA; AGEhIV Cohort Study Group. Multivariate normative comparison, a novel method for more reliably detecting cognitive impairment in HIV infection. AIDS. 2015 Mar 13;29(5):547-57. doi: 10.1097/QAD.0000000000000573. PMID 25587908
- [Result] Schouten J, Wit FW, Stolte IG, Kootstra NA, van der Valk M, Geerlings SE, Prins M, Reiss P; AGEhIV Cohort Study Group. Cross-sectional comparison of the prevalence of age-associated comorbidities and their risk factors between HIV-infected and uninfected individuals: the AGEhIV cohort study. Clin Infect Dis. 2014 Dec 15;59(12):1787-97. doi: 10.1093/cid/ciu701. Epub 2014 Sep 2. PMID 25182245
- [Result] Kooij KW, Wit FW, Bisschop PH, Schouten J, Stolte IG, Prins M, van der Valk M, Prins JM, van Eck-Smit BL, Lips P, Reiss P; AGEhIV Cohort Study group. Low bone mineral density in patients with well-suppressed HIV infection: association with body weight, smoking, and prior advanced HIV disease. J Infect Dis. 2015 Feb 15;211(4):539-48. doi: 10.1093/infdis/jiu499. Epub 2014 Sep 1. PMID 25180239
- [Derived] Vanbellinghen MC, Boyd A, Kootstra NA, Schim van der Loeff MF, van der Valk M, Reiss P; AGEhIV Cohort study group. A Biomarker Profile Reflective of Preserved Thymic Function Is Associated With Reduced Comorbidities in Aging People With HIV: An AGEhIV Cohort Analysis. J Infect Dis. 2025 Mar 17;231(3):622-632. doi: 10.1093/infdis/jiae603. PMID 39658325
- [Derived] Verburgh ML, Boyd A, Schim van der Loeff MF, Bakker M, Wit FWNM, van der Valk M, Grobben M, van Pul L, Tejjani K, van Rijswijk J, van Gils MJ, Kootstra NA, van der Hoek L, Reiss P; AGEhIV Cohort Study. Similar Limited Protection Against Severe Acute Respiratory Syndrome Coronavirus 2 Omicron Infection in Vaccinated Individuals With HIV and Comparable Controls. Open Forum Infect Dis. 2024 Jul 8;11(7):ofae380. doi: 10.1093/ofid/ofae380. eCollection 2024 Jul. PMID 39070044
- [Derived] Verburgh ML, van der Valk M, Rijnders BJA, Reiss P, Wit FWNM. No association between use of tenofovir disoproxil fumarate, etravirine, or integrase-strand transfer inhibitors and acquisition or severe outcomes of SARS-CoV-2 infection in people with HIV in the Netherlands. AIDS. 2023 Jul 15;37(9):1481-1486. doi: 10.1097/QAD.0000000000003577. Epub 2023 Apr 13. PMID 37395254
- [Derived] Schaaf REA, Verburgh ML, Boyd A, Wit FW, Nieuwkerk PT, Schim van der Loeff MF, Reiss P; AGEhIV Study Group. Change in Substance Use and the Effects of Social Distancing on Health-Related Quality of Life and Depressive Symptoms During the COVID-19 Pandemic in People Living With and Without HIV. J Acquir Immune Defic Syndr. 2022 Nov 1;91(3):261-268. doi: 10.1097/QAI.0000000000003055. Epub 2022 Jul 13. PMID 36252241
- [Derived] Verboeket SO, Boyd A, Wit FW, Verheij E, Schim van der Loeff MF, Kootstra N, van der Valk M, van Steenwijk RP, Drummond MB, Kirk GD, Reiss P; AGEhIV Cohort Study. Changes in lung function among treated HIV-positive and HIV-negative individuals: analysis of the prospective AGEhIV cohort study. Lancet Healthy Longev. 2021 Apr;2(4):e202-e211. doi: 10.1016/S2666-7568(21)00033-7. PMID 36098121
- [Derived] Verburgh ML, Boyd A, Wit FWNM, Schim van der Loeff MF, van der Valk M, Bakker M, Kootstra NA, van der Hoek L, Reiss P. Similar Risk of Severe Acute Respiratory Syndrome Coronavirus 2 Infection and Similar Nucleocapsid Antibody Levels in People With Well-Controlled Human Immunodeficiency Virus (HIV) and a Comparable Cohort of People Without HIV. J Infect Dis. 2022 Jun 1;225(11):1937-1947. doi: 10.1093/infdis/jiab616. PMID 34929034
- [Derived] Verheij E, Kirk GD, Wit FW, van Zoest RA, Verboeket SO, Lemkes BA, Schim van der Loeff MF, Reiss P; AGEhIV Cohort. Frailty Is Associated With Mortality and Incident Comorbidity Among Middle-Aged Human Immunodeficiency Virus (HIV)-Positive and HIV-Negative Participants. J Infect Dis. 2020 Aug 17;222(6):919-928. doi: 10.1093/infdis/jiaa010. PMID 31956893
- [Derived] Verboeket SO, Wit FW, Kirk GD, Drummond MB, van Steenwijk RP, van Zoest RA, Nellen JF, Schim van der Loeff MF, Reiss P; AGEhIV Study Group. Reduced Forced Vital Capacity Among Human Immunodeficiency Virus-Infected Middle-Aged Individuals. J Infect Dis. 2019 Apr 8;219(8):1274-1284. doi: 10.1093/infdis/jiy653. PMID 30418599